CLINICAL TRIAL: NCT00902928
Title: A Randomized, Double-Blind, Double-Dummy, Parallel Group Study to Compare YM150 Bid and qd Doses and Enoxaparin for Prevention of Venous Thromboembolism in Subjects Undergoing Elective Hip Replacement Surgery
Brief Title: A Study Evaluating Efficacy and Safety of YM150 Compared to Enoxaparin in Subjects Undergoing Hip Replacement Surgery
Acronym: ONYX-3
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Europe B.V. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 150-CL-040; 2008-004416-13 (EudraCT Number)
Record Dates: First submitted 2009-04-30; First posted 2009-05-15 (Estimated); Last update posted 2015-10-27 (Estimated); Status verified 2015-10

CONDITIONS: Venous Thromboembolism; Arthroplasty, Replacement, Hip
Keywords: Elective hip replacement surgery; Factor Xa; Venous Thromboembolism; Thrombosis; Anticoagulants; Prevention; YM150
MeSH Terms: conditions — Venous Thromboembolism; Thrombosis | interventions — Enoxaparin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 1. YM150, Dose X, twice daily (Experimental)
  Interventions: Drug: YM150
- 2, YM150, Dose X, once daily (Experimental)
  Interventions: Drug: YM150
- 3. YM150, Dose Y, twice daily (Experimental)
  Interventions: Drug: YM150
- 4. YM150, Dose Y, once daily (Experimental)
  Interventions: Drug: YM150
- 5. Enoxaparin (Active Comparator)
  Interventions: Drug: enoxaparin

INTERVENTIONS:
Drug: YM150 — oral
  Arms: 1. YM150, Dose X, twice daily; 2, YM150, Dose X, once daily; 3. YM150, Dose Y, twice daily; 4. YM150, Dose Y, once daily
Drug: enoxaparin — SC injection
  Arms: 5. Enoxaparin

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of various doses of YM150 (the experimental drug) compared to enoxaparin in the prevention of venous thromboembolism in patients that are undergoing elective hip replacement surgery.

ELIGIBILITY:
Inclusion Criteria:

* Subject is scheduled for elective hip replacement surgery

Exclusion Criteria:

* Subject has active bleeding or any condition associated with increased risk of bleeding
* Subject has had major trauma or surgery within 3 months before planned hip replacement surgery or requires major surgery or other invasive procedures with potential for uncontrolled bleeding during the study
* Subject has had an MI or stroke within 3 months before planned hip replacement surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1992 (Actual)
Dates: Start 2009-04; Primary Completion 2010-06 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Incidence of symptomatic Venous Thromboembolisms and death from all causes | 12 days

SECONDARY OUTCOMES:
Incidence of all Venous Thromboembolic events | Until day 12, during the treatment period, follow-up period and entire study period
Incidence of Bleeding events | During the treatment period, follow-up period and entire study period

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Europe B.V.
Locations (145):
- United States (17):
  - Phoenix, Arizona
  - Tuscon, Arizona
  - Little Rock, Arkansas
  - Long Beach, California
  - Torrance, California
  - Aurora, Colorado
  - DeLand, Florida
  - Pinellas Park, Florida
  - Sarasota, Florida
  - Tamarac, Florida
  - Meridian, Idaho
  - Lexington, Kentucky
  - Baltimore, Maryland
  - Charleston, South Carolina
  - Austin, Texas
  - Dallas, Texas
  - Houston, Texas
- Australia (5):
  - Box Hill, Victoria
  - Ringwood East, Victoria
  - Windsor, Victoria
  - Perth, Western Australia
  - Kogarah
- Austria (4):
  - Graz
  - Innsbruck
  - Linz
  - Vienna
- Foča, Bosnia and Herzegovina
- Brazil (3):
  - Curitiba, Puerto Rico
  - Porto Alegre, Rio Grande do Sul
  - São Paulo, So Paulo
- Canada (6):
  - Red Deer, Alberta
  - Burlington, Ontario
  - Guelph, Ontario
  - Newmarket, Ontario
  - Thunder Bay, Ontario
  - Waterloo, Ontario
- Colombia (4):
  - Medellín, Antioquia
  - Bogota, Cundinamarca
  - Floridablanca, Santander Department
  - Barranquilla
- Czechia (9):
  - Brno
  - Chomutov
  - Havlíčkův Brod
  - Jihlava
  - Jindřichův Hradec
  - Klatovy
  - Liberec
  - Prague
  - Třebíč
- Denmark (5):
  - Copenhagen
  - Frederiksberg
  - Herlev
  - Hørsholm
  - Silkeborg
- Estonia (3):
  - Kohtla-Järve
  - Tallinn
  - Tartu
- Finland (2):
  - Jyväskylä
  - Oulu
- Germany (2):
  - Mainz
  - Marburg
- Hungary (8):
  - Budapest
  - Debrecen
  - Győr
  - Kecskemét
  - Szeged
  - Szekszárd
  - Székesfehérvár
  - Szolnok
- India (11):
  - Hyderabaad, Andhra Pradesh
  - Secunderabad, Andhra Pradesh
  - Secunderabad, Andhra Prasdesh
  - Vadodara, Gujarat
  - Gurgaon, Haryana
  - Jamshedpur, Jharkhand
  - Bangalore, Karnataka
  - Kormangala, Karnataka
  - Mangalore, Karnataka
  - Bhopal, Madhya Pradesh
  - Jaipur, Rajasthan
- Israel (5):
  - Afula
  - Haifa
  - Kfar Saba
  - Petah Tikva
  - Rehovot
- Italy (2):
  - Bologna
  - Milan
- Latvia (4):
  - Daugavpils
  - Liepāja
  - Riga
  - Valmiera
- Lithuania (3):
  - Kaunas
  - Klaipėda
  - Vilnius
- Norway (5):
  - Gjøvik
  - Kongsvinger
  - Lillehammer
  - Tynset
  - Tønsberg
- Poland (9):
  - Gmina Końskie
  - Głogów Małopolski
  - Krakow
  - Lodz
  - Lublin
  - Opole
  - Otwock
  - Poznan
  - Warsaw
- Romania (5):
  - Timișoara, Timiș County
  - Bucharest
  - Cluj-Napoca
  - Craiova
  - Iași
- Russia (8):
  - Kazan'
  - Moscow
  - Nizhny Novgorod
  - Novosibirsk
  - Omsk
  - Saint Petersburg
  - Samara
  - Yaroslavl
- Slovakia (3):
  - Banska Bysterica
  - Kosice Saca
  - Prešov
- South Africa (5):
  - Worcester, Cape Town
  - Benoni
  - Bryanston
  - Port Elizabeth
  - Pretoria
- Spain (4):
  - Barcelona
  - Castelló
  - Madrid
  - Palma Mallorca
- Sweden (5):
  - Kalmar
  - Motala
  - Mölndal
  - Stockholm
  - Varberg
- Ukraine (4):
  - Cherkassy
  - Ivano-Frankivsk
  - Lviv
  - Sevastopol
- United Kingdom (3):
  - Epsom, Surrey
  - London
  - Northampton

REFERENCES:
- [Derived] Eriksson BI, Agnelli G, Gallus AS, Lassen MR, Prins MH, Renfurm RW, Kashiwa M, Turpie AG. Darexaban (YM150) versus enoxaparin for the prevention of venous thromboembolism after total hip arthroplasty: a randomised phase IIb dose confirmation study (ONYX-3). Thromb Haemost. 2014 Feb;111(2):213-25. doi: 10.1160/TH13-04-0296. Epub 2013 Oct 17. PMID 24136153